CLINICAL TRIAL: NCT03909737
Title: Sauver Avec l'Azithromycine en Traitant Les Femmes Enceintes et Les Enfants (SANTE)
Brief Title: Oral Azithromycin to Prevent Stillbirths and Infant Mortality in Mali
Acronym: SANTE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Karen Kotloff, Professor and Head, Division of Infectious Disease and Tropical Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00084242
Record Dates: First submitted 2019-02-26; First posted 2019-04-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Stillbirths and Infant Mortality
MeSH Terms: conditions — Stillbirth; Infant Death

STUDY DESIGN:
Intervention Model Description: This study will enroll three study cohorts: (1) a rural cohort of pregnant mother-infant pairs based in the southern region of Sikasso where infant mortality rates are higher than the national average (2) a rural cohort of only infants enrolled from the same communities as the mother-infant pairs, and (3) an urban cohort of pregnant mother-infant pairs based in Bamako. Cohort 1 will use a 2x2 factorial design. The pregnant women will be randomized to receive either oral azithromycin or placebo, and their infants, once born, will be separately randomized to receive either oral azithromycin or placebo. Cohorts 2 and 3 will use a parallel design. In Cohort 2, infants will be randomized to either azithromycin or placebo. In Cohort 3, mother-infant pairs will be randomized in tandem to either azithromycin or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Azithromycin to pregnant women and azithromycin to infants (Experimental): 2 gram oral dose of Azithromycin to pregnant women at their 2nd and 3rd trimester antenatal care visits and during delivery, plus 20 mg/kg to 1 gram oral dose of azithromycin to infants at 6 and 14 week Expanded Programme on Immunization (EPI) visits
  Interventions: Drug: Azithromycin to pregnant women; Drug: Azithromycin to infants
- Azithromycin to pregnant women and placebo to infants (Experimental): 2 gram oral dose of Azithromycin to pregnant women at their 2nd and 3rd trimester antenatal care visits and during delivery, plus oral placebo to infants at 6 and 14 week EPI visits
  Interventions: Drug: Azithromycin to pregnant women; Other: Placebo to infants
- Placebo to pregnant women and azithromycin to infants (Experimental): Oral placebo to pregnant women at their 2nd and 3rd trimester antenatal care visits and during delivery, plus 20 mg/kg to 1 gram oral dose of azithromycin to infants at 6 and 14 week EPI visits
  Interventions: Drug: Azithromycin to infants; Other: Placebo to pregnant women
- Placebo to pregnant women and placebo to infants (Placebo Comparator): Placebo to pregnant women at their 2nd and 3rd trimester antenatal care visits and during delivery, plus oral placebo to infants at 6 and 14 week EPI visits
  Interventions: Other: Placebo to pregnant women; Other: Placebo to infants
- No intervention to pregnant women and azithromycin to infants (Experimental): No intervention to pregnant women and 20 mg/kg to 1 gram oral dose of azithromycin to infants at 6 and 14 week EPI visits
  Interventions: Drug: Azithromycin to infants; Other: No intervention to pregnant women
- No intervention to pregnant women and Placebo to infants (Placebo Comparator): No intervention to pregnant women and placebo to infants at 6 and 14 week EPI visits
  Interventions: Other: Placebo to infants; Other: No intervention to pregnant women

INTERVENTIONS:
Drug: Azithromycin to pregnant women — Azithromycin to pregnant women at antenatal care visits and during delivery
  Arms: Azithromycin to pregnant women and azithromycin to infants; Azithromycin to pregnant women and placebo to infants
Drug: Azithromycin to infants — Azithromycin to infants at 6 and 14 week EPI visits
  Arms: Azithromycin to pregnant women and azithromycin to infants; No intervention to pregnant women and azithromycin to infants; Placebo to pregnant women and azithromycin to infants
Other: Placebo to pregnant women — Placebo to pregnant women at antenatal care visits and during delivery
  Arms: Placebo to pregnant women and azithromycin to infants; Placebo to pregnant women and placebo to infants
Other: Placebo to infants — Placebo to infants at 6 and 14 week EPI visits
  Arms: Azithromycin to pregnant women and placebo to infants; No intervention to pregnant women and Placebo to infants; Placebo to pregnant women and placebo to infants
Other: No intervention to pregnant women — No intervention to pregnant women
  Arms: No intervention to pregnant women and Placebo to infants; No intervention to pregnant women and azithromycin to infants

SUMMARY:
The double blind randomized controlled trial will assess the efficacy of oral azithromycin administered to pregnant women and/or infants during routine care in preventing stillbirths and mortality through 6-12 months of age in Mali, West Africa, where rates of infant and under five mortality are among the highest in the world.

DETAILED DESCRIPTION:
This trial will assess the efficacy of oral azithromycin given during routine health care visits in preventing stillbirths and mortality through 6-12 months of age in Mali, West Africa, where rates of infant and under five mortality are among the highest in the world. Using an individually randomized placebo-controlled double-masked trial design, pregnant women will receive a single dose of oral azithromycin or placebo at their second and/or third trimester antenatal care visits and during labor, and to infants at their DPT-1 and DPT-3 vaccination visits, which occur at approximately 6 and 14 weeks of age, respectively. The two co-primary outcomes are (1A) a composite outcome of stillbirths and mortality through 6-12 months of age and (1B) mortality between 6 weeks and 6-12 months of age. The study sample size is powered to detect a 20% relative reduction in both of the two co-primary outcomes. The study is designed to inform policymakers regarding the effectiveness of azithromycin for the prevention of stillbirth and infant mortality in both urban and rural parts of the country when administered during routine antenatal and intrapartum care and infant immunization visits. To achieve this aim, three cohorts will be enrolled: a mother-infant cohort in a rural part of the country with infant mortality rates that are higher than the national average, a supplemental infant-only cohort enrolled form the same rural communities, and third urban mother-infant cohort residing in Bamako, Mali's capital. Sub studies designed to elucidate the protective mechanisms of azithromycin treatment will be embedded within the larger study and will be added in the future.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women:

1. Participant is attending an ANC visit between 13 and 37 weeks gestation, with gestational age estimated using fundal height measurements and/or maternal report of quickening, at a participating health facility.
2. Participant is able to understand and comply with planned study procedures.
3. Participant has provided informed consent prior to initiation of any study procedures.
4. Participant intends to reside in the study area until her newborn infant is at least 12 months old.

Infants:

Enrollment of pregnant women and their unborn infants will happen simultaneously. Infants attending routine immunization visits at eligible health facilities whose mothers were not enrolled in the study will be eligible for enrollment in the supplemental infant cohort within the rural study cohort with the following inclusion criteria:

1. Infant is <12 mo attending a DTP-1 routine vaccination visit at a participating health facility.
2. Parent or guardian is able to understand and comply with planned study procedures.
3. Parent or guardian has provided informed consent prior to initiation of any study procedures.
4. Parent or guardian intends to reside in the study area until participant is at least 12 months old.

Exclusion Criteria:

1. Allergy to macrolides or azalides.
2. Any condition that, in the opinion of the investigator, might compromise the well-being of the participant or compliance with study procedures.
3. Medical treatment that requires administration of azithromycin (this can be a temporary exclusion if the drug is later discontinued).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99700 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of stillbirths and infant mortality through 6-12 months of age | 6 to 12 months
  Delivery outcomes assessed at intrapartum study visit and infant vital status assessed at 6 and 12 month study visits.
Rate of infant mortality between 6 weeks and 12 months of age | 6 weeks to 12 months
  Infant vital status will be assessed at 6 and 12 month study visits.

SECONDARY OUTCOMES:
Gestational age at birth | 3-6 months
  Gestational age will be estimated at enrollment and at delivery.
Birth weight | 3-6 months
  Birth weight will be measured.
The incremental cost-effectiveness ratio of adding azithromycin to standard of care in Mali | 6 to 18 months
  Costs associated with the delivery of azithromycin will be measured and the cost-effectiveness ratio will be estimated using efficacy data from the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Kotloff, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Centre pour le Developpement des Vaccins - Mali, Bamako, Mali

REFERENCES:
- [Derived] Driscoll AJ, Haidara FC, Tapia MD, Deichsel EL, Samake OS, Bocoum T, Bailey JA, Fitzpatrick MC, Goldenberg RL, Kodio M, Moulton LH, Nasrin D, Onwuchekwa U, Shaffer AM, Sow SO, Kotloff KL. Antenatal, intrapartum and infant azithromycin to prevent stillbirths and infant deaths: study protocol for SANTE, a 2x2 factorial randomised controlled trial in Mali. BMJ Open. 2023 Aug 30;13(8):e067581. doi: 10.1136/bmjopen-2022-067581. PMID 37648393